CLINICAL TRIAL: NCT05615701
Title: Image Quality of the EOSedge Radiographic System Versus a Standard Digital Radiographic (DR) System for Preoperative Assessment for Hip Replacement or Revision Surgery
Brief Title: Image Quality of EOSedge for Radiographic Evaluation of Hip Implant
Acronym: PreHIPEOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sufficient number of subjects included for analyzes
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL22_0298
Record Dates: First submitted 2022-10-27; First posted 2022-11-14 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Hip Osteoarthritis; Hip Prosthesis Infection
Keywords: EOS; Radiography; Hip; Hip replacement; Image quality
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EOSedge imaging (Other): Single arm study : All subjects include in the study underwent micro-dose EOS x-ray and digital radiography for radiographic evaluation of hip implant
  Interventions: Diagnostic Test: EOSedge imaging

INTERVENTIONS:
Diagnostic Test: EOSedge imaging — Hip X-ray evaluation in an EOSedge imaging for preoperative assessment for hip replacement or revision surgery

SUMMARY:
EOSedge is a precise, low dose imaging system that delivers full body, high-quality images covering the full set of musculoskeletal and orthopedic exams.

The objective of the study is to evaluate the quality of the focused pelvis/hip X-ray images on EOSedge compared to those performed on DR (current practice) to perform a preoperative radiographic evaluation of hip implant, A sufficient image quality on focused X-ray images performed on EOSedge would allow (1) to avoid the passage on two different radiographic systems (saving time) (2) to reduce the patient's x-ray radiation dose

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older
* Came to the imaging department to perform a preoperative assessment for hip replacement or revision

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient participating in an interventional study
* Patient unable to read and/or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Score of Image quality | Day 0
  Each criteria is quantitative and combined to obtain a final quantitative score :
  * Perfect reproduction = 2 / Moderate reproduction = 1 / Poor or uninterpretable reproduction = 0
  * Artifacts ? = no or absence of periprosthetic material = 1; YES = 0
  * X-ray image acceptable ? = Fully acceptable = 2; Acceptable only under limited clinical conditions = 1; Unacceptable (indicate why) = 0; OUTOCOME = FINAL SCORE
    1. European C, Directorate-General for R, Innovation, Carmichael J, Moores B, Maccia C. Guide européen relatif aux critères de qualité des clichés de radiodiagnostic: Publications Office, 2000.
    2. Kogon PL, Lumsden R. How do you critique your radiographs? The Journal of the Canadian Chiropractic Association. 1993; 37(4):230-232.
    3. Cook JV, Kyriou JC, Pettet A, Fitzgerald MC, Shah K, Pablot SM. Key factors in the optimization of paediatric X-ray practice. The British journal of radiology. 2001; 74(887):1032-1040.

SECONDARY OUTCOMES:
Dosimetry | Day 0
  The X-ray exposure dose induced by standard radiography and EOSedge will be compared.
  The radiation delivered to the patient during standard and EOSedge radiography will be quantified according to the dose × area product (DAP) [Gy.cm2] (dose * area product), for each exposure
Dosimetry | Day 0
  The X-ray exposure dose induced by standard radiography and EOSedge will be compared.
  The radiation delivered to the patient during standard and EOSedge radiography will be quantified according to the entry dose [mGy]

CONTACTS AND LOCATIONS:
Overall Officials: Catherine c-cyteval@chu-montpellier.fr, MD, PhD, Principal Investigator — Departement of Medical Imaging - Montpellier University hospital LAPEYRONIE Hospital
Locations (1):
- Departement of Medical Imaging, Montpellier, Occitanie, France